CLINICAL TRIAL: NCT03173755
Title: Relationships of Pain, Discomfort and Enjoyment During Exercise to Weight Status and Diet Quality.
Brief Title: Pain Discomfort Enjoyment Levels During Moderate Exercise
Status: Completed | Type: Observational
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Martin Binks, Associate Professor, Texas Tech University
Other Study IDs: TTUIRB2017-247
Record Dates: First submitted 2017-05-26; First posted 2017-06-02 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with normal weight
- people with overweight and obesity

SUMMARY:
In order to better understand how pre-existing pain and also discomfort/enjoyment during exercise may influence physical activity and be related to body weight the investigators are seeking to examine these as they relate to overweight/obesity compared to normal weight individuals. Ultimately, the investigators think that people with obesity may have more and be more sensitive to pain and have lower discomfort tolerance that may lead them to experience exercise more negatively. In the real world, this could result in them stopping exercise sooner or avoiding exercise all together. Therefore it is important for the investigators to begin to understand this issue better. In addition, some preliminary studies in animals suggest that the quality of the diet may influence pain sensitivity. This has yet to be examined in humans. As such the investigators will examine whether self-reported diet quality and also some markers in participants' blood that can tell the investigators about the recent quality of a person's diet, are related to the measures of pain, enjoyment and discomfort during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years.
* BMI ≥ 18.5 kg/m2.
* Typically exercise (moderate-intensity aerobic exercise - e.g. brisk walking) less than 150 minutes per week (last 3 months)
* No known contraindications for participating in up to 42 minutes of moderate intensity physical activity.
* Have not been told by a qualified healthcare provider to avoid moderate physical activity.

Exclusion Criteria:

* Unable/unwilling to provide informed consent.
* Having motor impairment.
* Currently diagnosed with diabetes mellitus, experiencing uncontrolled hypertension (i.e. systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) > 90 mmHg), having a history of ischemic heart disease, cerebrovascular accidents, neurological disease or current/past severe psychiatric illness (e.g. severe depression, psychosis, schizophrenia) that required hospitalization, severe current untreated depression (i.e. score in the severe depression range on the Hospital Anxiety and Depression Scale; HADS), current suicidal ideation, and current or past suicide attempts.
* Women who are pregnant or nursing.
* Diagnosed history of eating disorders such as bulimia nervosa, anorexia nervosa.
* Diagnosed history of substance abuse or alcohol abuse.
* Currently undergoing pain management treatment (pharmacologic and or behavioral).
* Currently taking anti-depressant medicines
* Have been instructed by a qualified healthcare provider to refrain from moderate physical activity at any time during the last 12 months (reasons other than minor orthopedic injury etc.).
* Any implanted medical devices (e.g. pacemaker).
* Currently smoking (within last 12 months).

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study will recruit participants from Lubbock Texas Community and surrounding regions.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of self-report measurement of pain (Short Form McGill Pain Questionnaire) according to BMI. | Baseline
  Comparison of self-report measurement of pain (Short Form McGill Pain Questionnaire) according to BMI (weight and height will be combined to report BMI in kg/m2).
Comparison of self-report measurement of pain (Subjective Pain Rating Scale) according to BMI. | Baseline
  Comparison of self-report measurement of pain (Subjective Pain Rating Scale) according to BMI (weight and height will be combined to report BMI in kg/m2).
Comparison of physical activity-induced pain (Subjective Pain Rating Scale) according to BMI. | minute zero through minute 42 of single exercise testing session (pre- post- session)
  Comparison of physical activity-induced pain (Subjective Pain Rating Scale) according to BMI (weight and height will be combined to report BMI in kg/m2).

SECONDARY OUTCOMES:
Comparison of self-report measurement of pain (Short Form McGill Pain Questionnaire) according to diet quality index. | Baseline
  Comparison of self-report measurement of pain (Short Form McGill Pain Questionnaire) according to diet quality index (DQI; is a factor analytically derived composite score of 5 nutritional quality biomarkers <plasma alkylresorcinol, Omega-3 index, serum fatty acid composition, serum carotenoids, and serum selenium>.)
Comparison of self-report measurement of pain (Subjective Pain Rating Scale) according to diet quality index. | Baseline
  Comparison of self-report measurement of pain (Subjective Pain Rating Scale) according to diet quality index (DQI is a factor analytically derived composite score of 5 nutritional quality biomarkers < plasma alkylresorcinol, Omega-3 index, serum fatty acid composition, serum carotenoids, and serum selenium>.)
Comparison of objectively measured pain tolerance (Dolorimetry) according to BMI. | Baseline
  Comparison of objectively measured pain tolerance (Dolorimetry) according to BMI (weight and height will be combined to report BMI in kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, PhD, Principal Investigator — Texas Tech University - Department of Nutritional Sciences
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States